CLINICAL TRIAL: NCT03475017
Title: Effects of Curcumin Supplementation in Inflammation, Oxidative Stress and Intestinal Microbiota in Patients With Chronic Kidney Disease
Brief Title: Effects of Curcumin in Patients in Chronic Kidney Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Denise Mafra (Other)
Responsible Party: Sponsor-Investigator, Denise Mafra, Doctor, Universidade Federal Fluminense
Organization: Universidade Federal Fluminense (Other)
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Health Services Research
Other Study IDs: Denisemafra4
Record Dates: First submitted 2018-02-21; First posted 2018-03-23 (Actual); Last update posted 2023-12-15 (Actual); Status verified 2023-12

CONDITIONS: Chronic Kidney Diseases
MeSH Terms: conditions — Renal Insufficiency, Chronic | interventions — Curcumin; piperine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Supplement A (Active Comparator): Administration of 3 capsules with 500mg of curcumin and piperine per day, for 12 weeks
  Interventions: Dietary Supplement: Active Comparator: Supplement A
- Supplement B (Placebo Comparator): Administration of 3 capsules with 500mg of placebo (maize starch) per day, for 12 weeks
  Interventions: Dietary Supplement: Placebo Comparator: Supplement B

INTERVENTIONS:
Dietary Supplement: Active Comparator: Supplement A — The patients will receive 3 capsules per day containing 500mg of curcumin and 5mg of piperine for 4 weeks
  Other Names: Curcumin and piperine
  Arms: Supplement A
Dietary Supplement: Placebo Comparator: Supplement B — The patients will receive 3 capsules of placebo per day containing 500mg of maize starch for 4 weeks
  Other Names: Placebo
  Arms: Supplement B

SUMMARY:
Many studies have been conducted to identify therapeutic strategies to modulate inflammation and oxidative stress, complications that contribute to the increased morbidity and cardiovascular mortality in patients with chronic kidney disease (CKD). Among several non-pharmacological strategies, the use of bioactive compounds has emerged as a potential approach to reduce these complications in CKD patients. In this context, turmeric/curcumin may have positive consequences in terms of cardiovascular and nephroprotection because of its antibacterial, antiviral, anti-inflammatory and anti-oxidative effects. The aim of this study is the role of curcumin as a nutritional strategy to reduce cardiovascular risk factors as inflammation and oxidative stress in CKD patients.

DETAILED DESCRIPTION:
This is a longitudinal study of the type randomized crossover, double-blind, placebo-controlled, washout period. We selected 30 patients with CKD in hemodialysis at Clínica Renalcor / RJ (second sample calculation, considering p = 0.05 and test power of 80%). Eligible patients of both genders, previously evaluated and authorized by the medical staff of the clinic, were invited to participate in the research.

The research was carried out after signing the free and informed consent form, according to the standards of the local Research Ethics Committees and required by Resolution 466 of December 12, 2012 (Conselho Nacional de Saúde), based on the guidelines of the Declaration of Helsinki and of the World Medical Association on human research. This project was approved by the Ethics Committee of the Faculty of Medicine / UFF, number: 2.346.933. It is registered with ClinicalTrials.gov under the number NCT 03475017.

Inclusion and exclusion criteria:

Patients with stage 5 CKD (GFR <15 mL / min) on hemodialysis for more than 6 months, aged at least 18 years, and who had arteriovenous fistula (AVF) as vascular access were included in the study. Patients who were pregnant, smokers, antibiotics in the last 3 months, antioxidant supplements and habitual turmeric and / or turmeric intake, besides those with autoimmune and infectious diseases, cancer, hepatic diseases and AIDS were not included in the study.

The food intake was evaluated at the beginning and at the end of the intervention through the 24-h food recall technique. The analysis of total energy intake (kcal/kg), carbohydrates (%), lipids (%), protein (g/kg), phosphorus (mg) and potassium (mg) were estimated using NutWin® software.

Assessment of nutritional status Patients had their body weight (kg), height (m), arm circumference (cm), waist circumference (WC) (cm) and skinfold measurements (mm) (biceps, triceps, subscapular, and suprailiac) measured with the aid of calibrated balance, stadiometer, tape measure and Lange Skinfold Caliper type adipometer (Cambridge Scientific Industries Inc.) before and after intervention. Body mass index (BMI) was calculated from dry body weight (kg) divided by squared height (m). Arm muscle area and body fat percentage were calculated. All measurements were performed after the dialysis session by a trained staff member.

Blood collection and biochemical analyzes Samples were collected in the morning after a 12-h fasting before dialysis and immediately after arteriovenous fistula puncture in Vacutainer® tubes containing ethylenediamine tetraacetic acid (EDTA) with anticoagulant (1.0 mg/mL). After collection, an aliquot was used for the analysis with whole blood and another one was centrifuged at 2500 rpm for 10 min at 4 C to obtain the plasma, which was distributed in 1.5 mL polypropylene eppendorfs tubes, identified and aliquoted for each analysis and stored at 80 C for further analysis. The whole blood was used to obtain the peripheral blood mononuclear cells (PBMC).

Real time PCR analysis Nrf2, NF-kB mRNA expression were evaluated from PBMC using quantitative real-time polymerase chain reaction (qPCR). TaqMan Gene Expression (Thermo Fisher®) assays for the detection of Nrf2 (Hs00975961_g1), NF-kB (Hs00765730_m1), and GAPDH (Hs02758991_g1) control mRNA expression were used. The Prism 7500 Sequence Detection System ABI (Applied Biosystems®) and the standard cyclic conditions were used for PCR amplification. NRf2, NF-kB mRNA expression were normalized against GAPDH, and the level of expressionwas calculated using the DDCT (delta delta threshold cycle) method.

Biochemical parameters Relevant information such as the etiology of CKD and age were collected from patients' records. Routine biochemical exams corresponding to collection dates, such as urea, Kt/v, hemoglobin and albumin, serum phosphorus, potassium, parathyroid hormone, glucose, and glycated hemoglobin were also obtained from routine medical records. Serum levels of high sensitivity C-reactive protein (hsCRP), total cholesterol, triglycerides, c-HDL were determined using BioClin® kits using the biochemical analyzer Bioclin BS-120 Chemistry Analyze. LDL was calculated using the Friedewald equation, considering triglyceride values below 400 mg/dL: LDL Cholesterol ¼ (Total Cholesterol) - (HDL Cholesterol) - (Triglycerides)/5.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of Chronic Kidney Disease
* Hemodialysis patients for more than 6 months
* Aged 18 years or older
* Must be able to swallow tablets

Exclusion Criteria:

* Patients pregnant
* Smokers
* Using antibiotics in the last 3 months
* Using antioxidant supplements in the last 3 months
* Usual intake of turmeric
* Usual intake Autoimmune
* Clinical diagnosis of infectious diseases
* Clinical diagnosis of Cancer
* Clinical diagnosis of AIDS

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2018-02-22 (Actual); Primary Completion 2021-04-29 (Actual); Study Completion 2021-12-30 (Actual)

PRIMARY OUTCOMES:
Antioxidants and anti-inflammatory biomarkers | 4 weeks
  Get blood samples to evaluate the supplementation effects in antioxidants biomarkers- nuclear receptor factor 2 (Nrf2), glutathioneperoxidase (GPx), heme oxygenase-1 (HO-1)
Inflammatory biomarkers | 4 weeks
  Get blood samples to evaluate the supplementation effects in inflammatory biomarkers- factor nuclear kappa B (NFkB), interleukin 6 (IL-6), tumor necrosis factor alpha (TNF-alpha)

CONTACTS AND LOCATIONS:
Locations (1):
- Denise Mafra, Rio de Janeiro, Rio de Janeiro, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Alvarenga L, Salarolli R, Cardozo LFMF, Santos RS, de Brito JS, Kemp JA, Reis D, de Paiva BR, Stenvinkel P, Lindholm B, Fouque D, Mafra D. Impact of curcumin supplementation on expression of inflammatory transcription factors in hemodialysis patients: A pilot randomized, double-blind, controlled study. Clin Nutr. 2020 Dec;39(12):3594-3600. doi: 10.1016/j.clnu.2020.03.007. Epub 2020 Mar 13. PMID 32204978